CLINICAL TRIAL: NCT04591769
Title: Cuff Pressure During Surgical Retractor Splay and Postoperative Voice Outcome After Anterior Cervical Spine Surgery: Comparison Between Tapered-shaped and Conventional Cylindrical-shaped Endotracheal Tube
Brief Title: Tracheal Tube Cuff Shape and Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Ya-Chun Chu, MD, PhD, Division of Neuroanesthesia, Department of Anesthesiology, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-10-002C
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Intubation, Intratracheal; Pain, Postoperative; Dysphonia
MeSH Terms: conditions — Pain, Postoperative; Dysphonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be intubated by an anesthesiologist who is aware of the grouping. After tracheal intubation is finished, the cuff is connected to the pressure monitor system and another blinded assessor will adjust and record the minimal volume that is required for sealing the tracheal tube-ventilator. The cuff pressure will be monitored and recorded all throughout the surgical period. A blinded assessor will follow up the patient after the surgery and do the voice analysis. Patients are unaware of the type of tracheal tube they used and will score subjectively for the sore throat and postoperative dysphonia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T(Tapered- shaped) (Experimental): Tracheal intubation using TaperedGuard Tracheal Tube
  Interventions: Device: Different tracheal tube cuff design
- Group C(Cylindrical-shaped) (Active Comparator): Tracheal intubation using Hi-Contour Tracheal Tube
  Interventions: Device: Different tracheal tube cuff design

INTERVENTIONS:
Device: Different tracheal tube cuff design — Comparison of effect between 2 different designs of tracheal tube cuff

SUMMARY:
This is a randomized controlled trial focusing on the effect of different tracheal tube cuff shape; the tapered-shaped tracheal tube cuff versus the cylindrical-shaped tracheal cuff in anterior cervical spine surgery.

DETAILED DESCRIPTION:
High endotracheal cuff pressure (ETCP) during surgical retractor splay associates with recurrent laryngeal nerve paresis/ palsy and results in post-anterior cervical spine surgery (post-ACSS) dysphonia. Control of intraoperative ETCP during ACSS may benefit voice outcome. The taper-shaped tracheal tube cuff was originally designed as a new strategy to reduce fluid leakage across the conventional cylindrical cuff and prevention of ventilator associated pneumonia. Literature has revealed the just seal pressure for the tapered-shaped tracheal tube (TT) cuff was lower than conventional cylindrical cuff. Therefore the investigators hypothesize that use of a tapered-shaped ET cuff during the surgery can lead to a lower ETCP during retractors splay and improve voice recovery after ACSS. In this study, 80 patients were randomized into 2 groups, to receive endotracheal intubation using TaperGuard tracheal tube (tapered- shaped cuff) or a conventional tracheal tube (a cylindrical cuff). The just seal pressure, intraoperative cuff pressure, and postoperative sore throat and voice outcome are recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Receiving elective anterior cervical spine surgery
* Right side approach

Exclusion Criteria:

* Unstable cervical spine (acute trauma history, or dislocation/ subluxation in image studies)
* Anticipated difficult airway
* Facial anomaly that may hinder facemask ventilation
* Preoperative hoarseness or vocal cord palsy regardless of etiology
* Re-operation of cervical spine surgery or left side approach
* BMI >35
* Operation field involved cervical spine C1 or C2
* Unwilling to sign the informed consent
* Unwilling to finish the study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Just seal tracheal tube cuff pressure | 1 minute after anesthesia and tracheal intubation
  Minimal tracheal tube cuff pressure that prevent leakage of the ventilator system
Tracheal tube cuff pressure on retractor splay | Intraoperative monitoring
  Cuff pressure when the retractors are set-up and removed

SECONDARY OUTCOMES:
Sore throat-NRS | preOP(operation) day 1, post OP 2 hours, day 1, 2, 3, 7
  Postoperative sore throat, Numeric Rating Scale(NRS) 0~10; 0=no sore throat; 10=maximal sore throat
Sore throat-VAS | preOP(operation) day 1, post OP 2 hours, day 1, 2, 3, 7
  Postoperative sore throat, Visual Analogue Scale (VAS) 0~10; 0=no sore throat; 10=maximal sore throat
Subjective dysphonia | preOP day 1, post OP 2 hours, day 1, 2, 3, 7
  Hoarseness; Pitch; Loudness (0= none; 1= mild; 2= severe); compared with baseline
Subjective dysphonia-GRBAS score | One day before operation, and post operation day 1
  GRBAS (Grade, Roughness, Breathiness, Asthenia, Strain) score (normal, slight, moderate, severe); compared with baseline
Subjective dysphonia- Voice Handicap Index-10(VHI-10) | One day before operation, and post operation day 7
  VHI-10 questionnaire (0 best~40 worst; >15 may be abnormal)
Objective dysphonia | One day before operation(baseline), and post operation day 1
  Software voice analysis; compared with baseline
Postoperative complication | After operation to post operation day 7
  Any postoperative complication related complication

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Chun Chu, MD, PhD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee. Proposals should be directed to yachunchu@gmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Li YS, Tan EC, Tsai YJ, Mandell MS, Huang SS, Chiang TY, Huang WC, Chang WK, Chu YC. A Tapered Cuff Tracheal Tube Decreases the Need for Cuff Pressure Adjustment After Surgical Retraction During Anterior Cervical Spine Surgery: A Randomized Controlled, Double-Blind Trial. Front Med (Lausanne). 2022 Jun 29;9:920726. doi: 10.3389/fmed.2022.920726. eCollection 2022. PMID 35847807